CLINICAL TRIAL: NCT04641936
Title: Urine Metabolomics and Proteomics Profiling to Predict the Responses and Adverse Events of Immuno-Oncology-based Therapy in Patients With Metastatic Urothelial Carcinoma
Brief Title: Urine Omics Predicting IO Therapy Responses in mUC Patients
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202010097RINC
Record Dates: First submitted 2020-11-18; First posted 2020-11-24 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Metastatic Urothelial Carcinoma
Keywords: urothelial carcinoma; biomarkers; clinical responses; IO-based therapies; metabolomics; proteomics; Urine
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: fresh urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: Training cohort will be recruited in the first 24 months of the study period to generate urine metabolomic and proteomic profiles as predictive and prognostic markers.
  Interventions: Other: No intervention required
- Cohort B: Validation cohort will be recruited in the next 36 months of the study period.
  Interventions: Other: No intervention required

INTERVENTIONS:
Other: No intervention required — No intervention required

SUMMARY:
The study aims to identify urinary metabolite and protein markers that can predict anti-tumor efficacy and adverse events in subjects receiving IO-based therapies for metastatic urothelial carcinoma.

DETAILED DESCRIPTION:
This is a multi-center single-arm translational study where patients with mUC who are about to receive pre-determined IO-based anti-tumor therapy will be invited to participate the study. After signing the approved informed consent, eligible and consenting subjects will donate their fresh urine samples for subsequent untargeted metabolomics and proteomics study via GS-MS/MS and/or LC-MS/MS to identify potential metabolite and protein markers that are able to predict efficacy and side effects of IO-based therapies. All subjects in the first-line, maintenance after 1st line, second-line, or subsequent lines of IO-based therapy will be invited and recruited, but those who have received any IO-based therapy before the study can NOT be recruited.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age > 20 years
* 2. Subjects diagnosed as metastatic urothelial carcinoma (mUC)
* 3. Subjects who are about to receive IO-based therapy
* 4. ECOG performance 0, 1, 2, and 3
* 5. Life expectancy 3 months
* 6. eGFR > 15 ml/min/1.73 m2 (Stage IV Chronic Kidney Disease or better)
* 7. Willing to sign the informed consent form

Exclusion Criteria:

* 1. Subjects NOT willing to sign the informed consent form
* 2. Subjects with active infection or active urinary tract infection, as shown by urinary WBC > 5/HPF
* 3. Subjects having co-existing other malignancies that need active treatment. Those with other malignancies that do not need active treatment are allowed to join the study.
* 4. Subjects taking any immune-modulating agents, including but not limited to corticosteroid, immune-suppressants, etc. at the discretion of recruiting investigators
* 5. Subjects who have taken any CPIs before. However, subjects who have received intravesical or intrapelvic BCG instillation are allowed to enroll.
* 6. Subjects who have received anti-FGFR therapy, enfortumab vedotin or other systemic therapies within 12 weeks of screening are not allowed. However, subjects who had a washout period of the above agents for >12 weeks are allowed to enroll. Subjects who have received or are receiving cytotoxic chemotherapy are allowed to join the study.

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced and metastatic UC patients who will receive IO-based therapy.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-12-17 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 7 years
Progression-free survival (PFS) | 7 years
Duration of response (DOR) | 7 years
Overall survival (OS) | 7 years
Adverse event of special interest (AESI) | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Yeong Shiau Pu, MD PhD, Principal Investigator — Department of Urology, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No